CLINICAL TRIAL: NCT03120845
Title: Incidence of Post-operative Pain After Single-visit Versus Two-visit Root Canal Treatment of Teeth With Necrotic Pulp and Apical Periodontitis
Brief Title: Incidence of Post-operative Pain After Single-visit Versus Two-visit Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jorge Paredes Vieyra (Other)
Responsible Party: Sponsor-Investigator, Jorge Paredes Vieyra, D.D.D., MsC, PhD, Universidad Autonoma de Baja California
Organization: Universidad Autonoma de Baja California (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Postop pain
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Post-operative Pain
Keywords: Pain,; one-visit; two visits
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Dental Implantation, Endosseous, Endodontic

STUDY DESIGN:
Intervention Model Description: Ibuprofen for post operative pain. after RCT in one visit
Who Masked: Participant
Masking Description: To compare incidence of post-operative pain and apical healing after single-visit versus two-visit root canal treatment of teeth with necrotic pulp and apical periodontitis. Each participant received a root canal treatment (RTC)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post operative Pain in one visit RCT (Experimental): One visit RCT Ibuprofen for Post operative pain. Take 400 mg every 6 hours, a week after.
  Interventions: Procedure: One visit RCT
- Post operative pain in two-visits RCT (Experimental): Two visits RCT Ibuprofen for Post operative pain. Take 400 mg every 6-8 hours, a week after.
  Interventions: Procedure: Post operative pain in two-visits RCT

INTERVENTIONS:
Procedure: One visit RCT — Root canal treatment in one vist
  Other Names: Endodontic therapy
  Arms: Post operative Pain in one visit RCT
Procedure: Post operative pain in two-visits RCT — Root canal treatment in Two visits
  Other Names: Endodontic Therapy
  Arms: Post operative pain in two-visits RCT

SUMMARY:
Aim :to compare incidence of post-operative pain and apical healing after single-visit versus two-visit root canal treatment of teeth with necrotic pulp and apical periodontitis.

DETAILED DESCRIPTION:
Aim to compare incidence of post-operative pain and apical healing after single-visit versus two-visit root canal treatment of teeth with necrotic pulp and apical periodontitis.

Methodology: All teeth of the one and two-visit group were asymptomatic (92) and symptomatic (18) with a diagnosis of pulp necrosis (RCT cases) determined by hot and cold sensitivity tests and radiographically all teeth showed a small and irregular radiolucency at the tooth apex. Working length was established with EAL and confirmed radiographically. Reciprocating files (VDW, Munich Germany) were used to complete root canal preparation. EDTA served as a lubricant.

ELIGIBILITY:
Inclusion Criteria:

1. The aims and requirements of the study were freely accepted;
2. Treatment was limited to patients in good health;
3. All teeth had nonvital pulps and apical periodontitis, with or without a sinus tract;
4. A negative response to hot and cold pulp sensitivity tests;
5. Presence of sufficient coronal tooth structure for rubber dam isolation;
6. No prior endodontic treatment on the involved tooth
7. No analgesics or antibiotics were used five days before the clinical procedures began.

Exclusion Criteria:

1. Patients who did not meet inclusion requirements;
2. Patients who did not provide authorization for participation;
3. Patients who were younger than 16 years old;
4. Patients who were pregnant;
5. Patients who were diabetic;
6. Patients with a positive history of antibiotic use within the past month;
7. Patients whose tooth had been previously accessed or endodontically treated;
8. Teeth with root resorption,
9. Immature/open apex, or a root canal in which patency of the apical foramen could not be established were all excluded from the study. Teeth with periodontal pockets deeper than 4 mm also were excluded of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-02-02; Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-26 (Actual)

PRIMARY OUTCOMES:
Post-operative pain in one visit | one week
  Pain intensity measure with general pain scale Each patient will recall a week to evaluate post operative pain

CONTACTS AND LOCATIONS:
Overall Officials: Miguel O Osuna, DDS, Study Chair — SECRETARIA DE SALUD

IPD SHARING:
Plan to Share IPD: Yes
Each participant will be evaluated a week after the treatment.

REFERENCES:
- [Background] Paredes-Vieyra J, Enriquez FJ. Success rate of single- versus two-visit root canal treatment of teeth with apical periodontitis: a randomized controlled trial. J Endod. 2012 Sep;38(9):1164-9. doi: 10.1016/j.joen.2012.05.021. Epub 2012 Jul 26. PMID 22892729